CLINICAL TRIAL: NCT05796089
Title: A Phase II Study of Platinum and Etoposide Chemotherapy, Durvalumab With Thoracic Radiotherapy in the First Line Treatment of Patients With Extensive-stage Small-cell Lung Cancer
Brief Title: Chemotherapy and Immunotherapy in Extensive-Stage Small-Cell Lung Cancer With Thoracic Radiotherapy
Acronym: CHEST RT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 20.01 CHEST RT
Record Dates: First submitted 2023-02-09; First posted 2023-04-03 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Extensive-Stage Small-Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Carboplatin; Cisplatin; Platinum; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Participants will receive Durvalumab concurrently with chemotherapy (etoposide with carboplatin or cisplatin) for 4 cycles.
  Interventions: Radiation: Thoracic Radiotherapy; Drug: Etoposide with Carboplatin or Cisplatin; Drug: Durvalumab

INTERVENTIONS:
Radiation: Thoracic Radiotherapy — Participants will receive thoracic radiotherapy to a dose of 30 Gray (Gy) in 10 fractions (3 Gy per day) concurrently with cycle 3 or 4 of chemo-immunotherapy (Group 1).
  Participants who are unsuitable for concurrent radiotherapy may receive consolidation radiotherapy. Consolidation thoracic radiotherapy will be administered to a dose of 30 Gy in 10 fractions, following 4 cycles of chemo-immunotherapy (Group 2).
  Treatment fractions will be delivered daily, where treatment should be completed within 15 days (9-10 fractions a fortnight).
  Other Names: Thoracic Radiation Therapy
Drug: Etoposide with Carboplatin or Cisplatin — The chemotherapy in this study is a standard treatment for extensive-stage small-cell lung cancer (EC-SCLC). The combination of chemotherapy (etoposide + carboplatin or etoposide + cisplatin) which the participant will receive is dependent on what is standard at the treatment centre.
  Chemotherapy will be administered via an intravenous infusion every 3 weeks (21 days) for 4 cycles.
  Other Names: Platinum + Etoposide; EP Chemotherapy
Drug: Durvalumab — The immunotherapy in this study is a standard treatment for ES-SCLC.
  Participants will receive a dose of 1500 mg of Durvalumab via an intravenous infusion every 3 weeks (21 days) for 4 cycles, concurrently with chemotherapy.
  A 1500 mg maintenance dose of Durvalumab will administered every 4 weeks after completion of chemotherapy (monotherapy).
  Other Names: IMFINZI; MEDI4736

SUMMARY:
This is a prospective, multi-centre, single arm, phase 2, open label clinical trial of patients with untreated extensive-stage small-cell lung cancer (ES-SCLC) suitable for first-line platinum-based chemotherapy. The aim of the trial is to assess safety, feasibility and describe efficacy of the addition of concurrent thoracic radiotherapy to usual treatment of chemotherapy and immunotherapy (durvalumab) in patients with ES-SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent
* Histologically or cytologically documented ES-ECLC
* Thoracic disease deemed suitable for radiation therapy following initial systemic therapy
* If brain metastases present, then they are to be;

  1. asymptomatic without steroid therapy may be included or
  2. have required treatment (radiotherapy and/or surgery) and are clinically stable and patient is on a stable or reducing steroid dose of no more than dexamethasone 4mg/day (or equivalent)
* Patients must be considered suitable to receive platinum-based chemotherapy regimen as first-line treatment for ES-SCLC
* ECOG performance-status score of 0 or 1 at registration
* Life expectancy ≥ 12 weeks at registration
* Body weight > 30 kg
* No prior exposure to immune-mediated therapy including, but not limited to, other anti-cytotoxic T-lymphocyte-associated antigen-4, anti-programmed cell death-1, anti-programmed cell death ligand-1, and anti-programmed cell death ligand-2 antibodies, excluding therapeutic anticancer vaccines
* Adequate organ and marrow function as defined in the Protocol
* Female patients who;

  1. are willing to use adequate contraceptive measures until 90 days after the final dose of trial treatment
  2. are not breast feeding
  3. have a negative pregnancy test prior at registration if of child bearing potential or have evidence of non-child bearing potential by fulfilling the criteria as stated in the Protocol at screening

Exclusion Criteria:

* Treatment with any of the following:

  1. Concurrent chemotherapy (not relevant to patients registered prior to cycle 2 who will have received a cycle of platinum/etoposide chemotherapy), investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
  2. An investigational product during the last 4 weeks
  3. High dose radiotherapy to the chest prior to systemic therapy precluding further thoracic radiation therapy. Radiation therapy outside of the chest for palliative care (i.e., bone metastasis) is allowed but must be completed before first dose of the trial medication
  4. Immunosuppressive medication within 14 days before the first dose of durvalumab. Some exceptions apply
  5. Live, attenuated vaccine within 30 days prior to the first dose of durvalumab
  6. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of Durvalumab. Surgical procedures to obtain a lung cancer diagnosis or for palliation are allowed
* Medical contraindication to, known allergy or hypersensitivity to durvalumab, etoposide, carboplatin (patients with allergy/hypersensitivity to carboplatin may receive cisplatin), cisplatin, or any of their excipients
* History of allogeneic organ transplantation
* Has a para-neoplastic syndrome (PNS) of autoimmune nature, requiring systemic treatment (systemic steroids or immunosuppressive agents) or has a clinical symptomatology suggesting worsening of PNS. Patients with hyponatraemia considered due to SIADH syndrome are eligible
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis. Some exceptions apply
* Interstitial lung disease/pulmonary fibrosis. Patients with emphysema and associated limited areas of pulmonary fibrosis are eligible
* Uncontrolled intercurrent illness
* History of another primary malignancy. Some exceptions apply
* History of leptomeningeal carcinomatosis
* History of active primary immunodeficiency
* Patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety of chemo-immunotherapy with concurrent thoracic radiotherapy | From date of consent to 90 days after trial treatment is discontinued
  Group 1 and Group 2 will be compared for the presence of toxicity, whereby the proportion of grade 3 or higher pneumonitis and grade 3 or higher oesophagitis will be monitored using the NCI Common Terminology Criteria for Adverse Events v5.
Feasibility of chemo-immunotherapy with concurrent thoracic radiotherapy | From date of consent to 90 days after trial treatment is discontinued
  Group 1 and Group 2 will be compared for the proportion of participants which received concurrent radiotherapy vs the proportion of participants which did not receive concurrent radiotherapy.
  The two groups will also be assessed by the proportion of participants in which discontinued thoracic radiotherapy.

SECONDARY OUTCOMES:
Overall Survival | 12 months
  Overall survival will be defined as the time from the Cycle 1 day 1 of chemotherapy until the date of death by any cause. Participants who are alive by the analysis time point will be censored at the trial close out date.
Progression free survival | 6 and 12 months
  Progression free survival will be defined as the time from Cycle 1 Day 1 of chemotherapy until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the participant withdraws from therapy or receives another anticancer therapy prior to progression. Participants who are alive or have not progressed by the analysis time point will be censored at the latest of the dates contributing to a particular overall visit assessment.
Patterns of failure | From date of registration until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 152 weeks
  Patterns of failure assessed by the proportion of patients with first site of failure in: Thoracic, Extra-thoracic or cranial sites, seen on imaging (CT/MRI) and assessed by iRECIST and/or RANO-BM criteria. The first site of treatment relapse will be collected and categorised as thoracic, extra-thoracic or cranial.
Time to local failure and local control | 6 and 12 months
  Time to thoracic local failure and proportion of participants with thoracic local control.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hau, Study Chair — Westmead/Blacktown Hospital; Sagun Parakh, Principal Investigator — Austin Health
Locations (8):
- Australia (8):
  - Westmead Hospital, Sydney, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - St. Vincent's Hospital, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria

REFERENCES:
- [Derived] Parakh S, Gee H, Lim A, Vinod S, Wheeler C, Rooney B, Montgomery R, Harden S, Moore M, Lehman M, Bettington C, Moodie T, Barber J, Schmidt L, Dizon J, Leigh L, Oldmeadow C, Mitchell P, Hau E. Platinum and etoposide chemotherapy, durvalumab with thoracic radiotherapy in the first-line treatment of patients with extensive-stage small-cell lung cancer: CHEST-RT (TROG 20.01) Trial - protocol for a phase II study. BMJ Open. 2025 Jul 7;15(7):e101571. doi: 10.1136/bmjopen-2025-101571. PMID 40623886